CLINICAL TRIAL: NCT02171065
Title: A Multicentre Prospective Natural History Study Using Multimodality Imaging in Patients With ACS- PROSPECT II (Natural History Study), Combined With a Randomized, Controlled, Intervention Study - PROSPECT ABSORB (Randomized Trial)
Brief Title: PROSPECT II & PROSPECT ABSORB - an Integrated Natural History Study and Randomized Trial.
Acronym: P2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Abbott Medical Devices (Industry); Infraredx (Industry); The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PROSPECT II & PROSPECT ABSORB
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: NIRS/IVUS; multimodality imaging; PROSPECT
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guideline Directed Medical Therapy (Sham Comparator): Guideline Directed Medical Therapy
  Interventions: Device: sham
- ABSORB BVS + Guideline Directed Medical Therapy (Active Comparator): ABSORB BVS + Guideline Directed Medical Therapy
  Interventions: Device: ABSORB BVS

INTERVENTIONS:
Device: sham
  Arms: Guideline Directed Medical Therapy
Device: ABSORB BVS
  Arms: ABSORB BVS + Guideline Directed Medical Therapy

SUMMARY:
The present study has two components, an overall prospective observational study using multimodality imaging (PROSPECT II) that will examine the natural history of patients with unstable atherosclerotic coronary artery disease with the specific goal to establish the utility of low-risk intracoronary imaging modalities, IVUS and NIRS, to identify plaques prone to future rupture and clinical events. The randomized PROSPECT ABSORB substudy will examine whether treatment of vulnerable plaques with the Absorb Bioresorbable vascular scaffold (BVS) plus GDMT safely increases the minimum lumen area (MLA) at 24 months compared with GDMT alone.

The cutoff for inclusion in PROSPECT ABSORB will be a site-determined PB ≥65% (rather than the 70% cutoff identified in the original PROSPECT analysis (Stone et al., New England Journal of Medicine, 2011(5)) to account for an observed tendency for sites to underestimate plaque burden during acute treatment of ACS patients. Nonetheless, in PROSPECT, a core laboratory determined PB ≥65% was also associated with a high (7.0%) rate of major adverse cardiac event (MACE) during 3-year follow-up, a rate which may be reduced with a bioresorbable scaffold.

DETAILED DESCRIPTION:
Methodology:

PROSPECT II: Multicenter, prospective, natural history study of troponin positive patients with acute coronary syndromes (ACS) examined with angiography and intended for PCI for the initial culprit lesion(s). Prior to PCI all target lesions (those lesions for which PCI is planned) will be examined (if possible) by IVUS/NIRS. After successful PCI of all flow-limiting lesions determined angiographically and/or by FFR/iFR intended to be treated (termed "culprit lesions," whether responsible for the original ACS or otherwise flow-limiting and requiring PCI for complete revascularization), intravascular ultrasound (IVUS), and intracoronary near infrared spectroscopy (NIRS) will be performed over a 6-10 cm length in all three coronary arteries with a combined IVUS/NIRS catheter. Clinical and register follow-up will identify all new coronary events, the origin of which will be determined by follow-up angiography when clinically indicated. These lesions will be identified and compared to the baseline examination at a central angiographic and IVUS/NIRS core laboratory, and adjudicated to have arisen from either originally treated culprit lesions or untreated "non-culprit lesions." This will allow determination of the baseline patient-related and lesion-related variables in culprit and non-culprit lesions that increase the risk for future unanticipated cardiovascular events.

PROSPECT ABSORB (Randomized Trial): Patients with angiographically non-obstructive lesions that are not intended to undergo PCI based on the current standard of care, and that are site-assessed by IVUS to have plaque burden of ≥65% (which has previously been shown in the first PROSPECT study to identify lesions at high risk of causing future coronary events despite their non-obstructive angiographic appearance) will be randomized (1:1) to treatment with ABSORB BVS + guideline directed medical therapy (GDMT) versus GDMT alone. All such randomized patients will undergo repeat angiography and IVUS/NIRS after 25 months of follow-up.

Patient enrollment and procedure overview:

PROSPECT II: Patients with a troponin positive ACS within the prior 4 weeks (STEMI >12 hours or NSTEMI) in whom coronary angiography is planned will be screened and asked to participate in the study. After informed consent has been obtained and prior to PCI, all target lesions (those lesions for which PCI is planned) will be examined (if possible) by IVUS/NIRS. If the patient is successfully treated with PCI of all intended culprit lesions without major procedural complication(s), all three coronary arteries will be examined with IVUS/NIRS. The IVUS results will be visible (unblinded) to the operator, but the NIRS data will be blinded. The patient will be considered formally enrolled in PROSPECT II only after PCI of all intended target culprit lesions has been successfully completed with no major complication(s), and after the study imaging catheter is passed out of the guide catheter into a coronary artery (n = approximately 900 patients). If a staged procedure is required to achieve revascularization of all intended lesions, the patient will not be enrolled until after the staged procedure has been performed without major procedural complication(s). Once enrolled, IVUS and NIRS will be performed over a 6-10 cm length in all three coronary arteries with a combined IVUS/NIRS catheter to assess both the treated culprit lesion(s) and long segments of the untreated coronary tree. Patient enrollment and 3-vessel IVUS and NIRS imaging may be performed either in the same procedure during which the culprit PCI lesion(s) are treated, or during a subsequent angiographic procedure as long as this occurs within 4 weeks of the initial ACS presentation, and after successful and uncomplicated treatment of all target lesions. If the imaging catheter passed into a coronary artery for imaging a non-culprit segment of the coronary tree and no non-culprit segment imaging data is obtained (e.g. the catheter fails and a second catheter is not used), the patient will be disenrolled (discontinued) from the study, and only be followed up for safety purposes for 30 days.

PROSPECT ABSORB: Patients in whom one or more lesions are identified with (a) an angiographically visually estimated diameter stenosis of <70%; (b) a visually estimated reference vessel diameter (RVD) of 2.5 - 4.0 mm; (c) a visually estimated lesion length ≤50 mm; d) a site determined IVUS PB ≥65%; and (e) is located at least 10 mm from a previous stent and at least 10 mm of intervening segment between the previous stent and the non-culprit lesion does not have PB >50% will be enrolled in the PROSPECT ABSORB trial and randomized 1:1 to treatment with ABSORB BVS + GDMT versus GDMT alone (n = approximately 300 patients, 150 patients in each group). For patients with multiple qualifying lesions, a single lesion will be selected for randomization prior to assignment to BVS + GDMT versus GDMT alone.

Study follow-up:

PROSPECT II (Natural History Study)

Clinical follow-up:

Patients will be followed in the Scandinavian quality registers (eg, SWEDEHEART). Patients will undergo follow-up through register data collection and by calls by study coordinators at 1 month (30 days), 6 months (180 days), 12 months, and 24 months, assessing MACE and safety parameters. MACE will be followed in all patients throughout the whole study period until last patient has been followed for 24 months. Patients will then undergo follow-up through register data collection at yearly intervals starting at 3 years and through 15 years. Additional phone follow-up to patients may also be performed.

PROSPECT ABSORB (Randomized Trial)

Clinical follow-up:

Patients will be followed in the Scandinavian quality registers (eg, SWEDEHEART). Patients will undergo follow-up through register data collection and by calls by study coordinators at 1 month (30 days), 6 months (180 days), 12 months, and 24 months. MACE will be followed in all patients throughout the whole study period until last patient has been followed for 24 months. Patients will then undergo follow-up through register data collection at yearly intervals starting at 3 years and through 15 years, with additional phone follow-up subject to Executive Committee approval.

Angiographic follow-up:

All patients randomized in PROSPECT-ABSORB will undergo routine angiographic and 3-vessel IVUS/NIRS follow-up at 25 months; ie, 1 month after the 24 month telephone follow-up. The 25 month angiogram may be performed within a window of between 24.5 months and 28 months after enrollment.

Note: 25-month angiographic follow-up will not be required in PROSPECT-ABSORB randomized patients who either a) have had scaffold thrombosis or in-scaffold restenosis (DS>50% as determined by the angiographic core laboratory) at any time point prior to 25 months, OR b) have had a repeat angiogram ≥12 months after enrollment and in whom IVUS/NIRS of the randomized target lesion was performed.

ELIGIBILITY:
PROSPECT II

Inclusion Criteria:

1. Troponin positive ACS (STEMI >12 h or NSTEMI) occurring within the prior 4 weeks of enrollment, with symptoms consistent with acute ischemia lasting >10 minutes, intended for angiography and Percutaneous Coronary Intervention (PCI) if appropriate.
2. Patient must have one-vessel, two-vessel or three-vessel disease in native coronary arteries requiring PCI.
3. Successful PCI

Exclusion Criteria:

1. Known estimated creatinine clearance <30 ml/min.
2. Cardiogenic shock, decompensated hypotension or heart failure requiring intubation, inotropes, intravenous diuretics or a hemodynamic support device.
3. Patient has a known hypersensitivity, allergy or contraindication to any of the following: aspirin, both heparin and bivalirudin, all 3 of clopidogrel, prasugrel and ticagrelor, or to contrast that cannot be adequately pre-medicated.
4. Refractory ventricular arrhythmias (e.g. ventricular tachycardia or fibrillation) requiring either intravenous pharmacologic treatment or defibrillation during the index PCI procedure.
5. Persistent acute conduction system disease requiring temporary pacemaker insertion during the index PCI procedure.
6. Prior Coronary Artery Bypass Graft (CABG) at any time or planned CABG.
7. PCI is required of the left main coronary artery, or a left main stenosis is present with a visually estimated angiographic Diameter Stenosis (DS) of >30%.
8. Angiographic evidence of severe calcification and/or marked tortuosity of the target (culprit) or a non-culprit vessel is present that would preclude the feasibility of safe imaging of at least the proximal 6 cm of all vessels.
9. The presence of a chronic total occlusion of a major epicardial coronary vessel that is not successfully recanalized during the PCI procedure, and thus would preclude intravascular imaging.

PROSPECT ABSORB

Inclusion Criteria:

if one or more eligible lesions are identified which meet all of the following angiographic criteria:

1. The lesion is a de novo lesion (may be located in either the target or non-target vessel)
2. The lesion has an angiographic diameter stenosis <70%, and is not intended for revascularization based on angiographic criteria and Fractional Flow Reserve/Instantaneous wave-free ratio (FFR/iFR).

   Note: FFR/iFR should be performed on all noncritical lesions of greater than 40% visually estimated angiographic stenosis that are candidates for the ABSORB substudy.
3. The lesion has a site-determined IVUS plaque burden in at least one frame ≥65%. Note: Such a lesion may or may not be angiographically evident; i.e. the visually estimated angiographic diameter stenosis may range between 0% - <70%.
4. The reference vessel diameter of an eligible lesion is ≥2.5 mm - ≤4.0 mm (visually estimated) capable of being treated with a 2.5 mm, 3.0 mm, or 3.5 mm diameter BVS.
5. The lesion length of an eligible lesion is ≤50 mm (visually estimated), capable of being treated by no more than two BVS (maximum length of each BVS 28 mm), allowing for 2 mm BVS overlap and 2 mm of "normal" reference segment treatment at each edge.
6. The lesion must be at least 10 mm from a previously implanted stent/scaffold and an intervening 10 mm segment must not have plaque burden (PB) >50%
7. A bifurcation lesion may be enrolled only if the side branch is a) ≤2.5 mm in reference vessel diameter, AND b) has either no lesion requiring treatment, or atherosclerotic disease limited to within 5 mm of its origin from the parent vessel such that the operator believes that the side branch can be successfully treated with balloon angioplasty only (without a stent). If a stent subsequently becomes necessary, only a metallic drug-eluting stent (DES) may be used to treat the side branch with a T-stent technique.
8. Randomization must occur immediately after the 3-vessel imaging run in the PROSPECT II protocol. If the patient randomizes to BVS, BVS placement must be performed immediately after randomization.

Exclusion Criteria:

1. The randomized lesion cannot be within 10 mm of a lesion previously treated by PCI .
2. The randomized lesion may not be in the left main coronary artery.
3. The randomized lesion may not be an ostial Left Anterior Descending Coronary Artery (LAD) or ostial Left Circumflex Coronary Artery (LCX) lesion (defined as within 3 mm of the left main coronary artery).
4. The randomized lesion may not be an ostial Right Coronary Artery (RCA) lesion (defined as within 3 mm of the aorto-ostium).
5. Angiographic evidence of severe calcification and/or marked tortuosity of the target vessel and/or lesion intended for randomization is present that would make it unlikely that the BVS could be advanced to or across the lesion or be adequately expanded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Erlinge, MD, PhD, Study Chair — Lund University
Locations (1):
- David Erlinge, Lund, Sweden

REFERENCES:
- [Derived] Thrane PG, Maeng M, Maehara A, Botker HE, Mintz GS, Kjoller-Hansen L, Engstrom T, Matsumura M, Kotinkaduwa LN, Frobert O, Persson J, Wiseth R, Larsen AI, Jensen LO, Nordrehaug JE, Bleie O, Held C, James SK, Ali ZA, Erlinge D, Stone GW. Nonculprit Vulnerable Plaques and Prognosis in Myocardial Infarction With Versus Without ST-Segment Elevation: A PROSPECT II Substudy. Circulation. 2025 Jun 24;151(25):1767-1779. doi: 10.1161/CIRCULATIONAHA.124.071980. Epub 2025 Jun 23. PMID 40549845
- [Derived] Erlinge D, Tsimikas S, Maeng M, Maehara A, Larsen AI, Engstrom T, Kjoller-Hansen L, Matsumura M, Ben-Yehuda O, Botker HE, Frobert O, Persson J, Wiseth R, Jensen LO, Nordrehaug JE, Trovik T, Jensen U, Bleie O, Omerovic E, James SK, Rylance R, Sharma T, Ali ZA, Stone GW. Lipoprotein(a), Cholesterol, Triglyceride Levels, and Vulnerable Coronary Plaques: A PROSPECT II Substudy. J Am Coll Cardiol. 2025 Jun 3;85(21):2011-2024. doi: 10.1016/j.jacc.2025.04.013. PMID 40436465
- [Derived] Frobert O, Stone GW, Larsen AI, Zhou Z, Kotinkaduwa LN, Engstrom T, Kjoller-Hansen L, Maeng M, Matsumura M, Ben-Yehuda O, Botker HE, Persson J, Wiseth R, Jensen LO, Nordrehaug JE, Trovik T, Jensen U, Bleie O, James SK, Ali ZA, Omerovic E, Erlinge D, Maehara A. Relationships of hsCRP to High-Risk Vulnerable Plaque After NSTEMI: Insights From the PROSPECT II Trial. JACC Cardiovasc Interv. 2025 May 26;18(10):1217-1228. doi: 10.1016/j.jcin.2025.01.440. Epub 2025 Apr 23. PMID 40272345
- [Derived] Arslani K, Engstrom T, Maeng M, Kjoller-Hansen L, Maehara A, Zhou Z, Ben-Yehuda O, Botker HE, Matsumura M, Mintz GS, Frobert O, Persson J, Wiseth R, Larsen AI, Jensen LO, Nordrehaug JE, Bleie O, Omerovic E, Held C, James SK, Ali ZA, Erlinge D, Stone GW. Association Between Physiological Significance and Vulnerable Plaque Characteristics in Patients With Myocardial Infarction: A Prospect II Substudy. JACC Cardiovasc Imaging. 2025 Jun;18(6):696-706. doi: 10.1016/j.jcmg.2024.11.002. Epub 2025 Feb 24. PMID 39998456
- [Derived] Kjoller-Hansen L, Maehara A, Kelbaek H, Matsumura M, Maeng M, Engstrom T, Frobert O, Persson J, Wiseth R, Larsen AI, Jensen LO, Nordrehaug JE, Omerovic E, Held C, James S, Mintz GS, Ali ZA, Stone GW, Erlinge D. Impact of Lipidic Plaque on In-Stent and Stent Edge-Related Events After PCI in Myocardial Infarction: A PROSPECT II Substudy. Circ Cardiovasc Interv. 2024 Oct;17(10):e014215. doi: 10.1161/CIRCINTERVENTIONS.124.014215. Epub 2024 Sep 25. PMID 39319453
- [Derived] Gyldenkerne C, Maeng M, Kjoller-Hansen L, Maehara A, Zhou Z, Ben-Yehuda O, Erik Botker H, Engstrom T, Matsumura M, Mintz GS, Frobert O, Persson J, Wiseth R, Larsen AI, Jensen LO, Nordrehaug JE, Bleie O, Omerovic E, Held C, James SK, Ali ZA, Rosen HC, Stone GW, Erlinge D. Coronary Artery Lesion Lipid Content and Plaque Burden in Diabetic and Nondiabetic Patients: PROSPECT II. Circulation. 2023 Feb 7;147(6):469-481. doi: 10.1161/CIRCULATIONAHA.122.061983. Epub 2022 Dec 16. PMID 36524476
- [Derived] Erlinge D, Maehara A, Ben-Yehuda O, Botker HE, Maeng M, Kjoller-Hansen L, Engstrom T, Matsumura M, Crowley A, Dressler O, Mintz GS, Frobert O, Persson J, Wiseth R, Larsen AI, Okkels Jensen L, Nordrehaug JE, Bleie O, Omerovic E, Held C, James SK, Ali ZA, Muller JE, Stone GW; PROSPECT II Investigators. Identification of vulnerable plaques and patients by intracoronary near-infrared spectroscopy and ultrasound (PROSPECT II): a prospective natural history study. Lancet. 2021 Mar 13;397(10278):985-995. doi: 10.1016/S0140-6736(21)00249-X. PMID 33714389
- [Derived] Stone GW, Maehara A, Ali ZA, Held C, Matsumura M, Kjoller-Hansen L, Botker HE, Maeng M, Engstrom T, Wiseth R, Persson J, Trovik T, Jensen U, James SK, Mintz GS, Dressler O, Crowley A, Ben-Yehuda O, Erlinge D; PROSPECT ABSORB Investigators. Percutaneous Coronary Intervention for Vulnerable Coronary Atherosclerotic Plaque. J Am Coll Cardiol. 2020 Nov 17;76(20):2289-2301. doi: 10.1016/j.jacc.2020.09.547. Epub 2020 Oct 15. PMID 33069847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 10, 2014, and December 20, 2017, 902 patients at 16 sites were enrolled in PROSPECT II.
Pre-assignment Details: Four patients were disenrolled because non-culprit lesion imaging were not acquired. Among the rest of 898 patients, 182 patients with angiographically nonobstructive lesion but with plaque burden>=65% were enrolled in PROSPECT-ABSORB, and randomized to Absorb-bioresorbable vascular scaffold (BVS) plus guideline-directed medical therapy (GDMT) (n=93) versus GDMT alone (n=89).
Groups:
- Guideline Directed Medical Therapy in PROSPECT-ABSORB and PROSPECT II: Patients were enrolled in PROSPECT-ABSORB and randomized to guideline-directed medical therapy (GDMT) group. Patients remain in PROSPECT II cohort.
- ABSORB BVS + GDMT in PROSPECT-ABSORB and PROSPECT II: Patients were enrolled in PROSPECT-ABSORB and randomized to ABSORB-BVS + GDMT group. Patients remain in PROSPECT II cohort.
- PROSPECT II Only: Patients were not enrolled in PROSPECT-ABSORB. Patients remain in PROSPECT II.
Period: Overall Study
Arm/Group | Guideline Directed Medical Therapy in PROSPECT-ABSORB and PROSPECT II | ABSORB BVS + GDMT in PROSPECT-ABSORB and PROSPECT II | PROSPECT II Only
Started | 89 | 93 | 716
Completed | 88 | 93 | 715
Not Completed | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Guideline Directed Medical Therapy (GDMT) in PROSPECT-ABSORB and PROSPECT II: Patients were enrolled in PROSPECT-ABSORB and randomized to GDMT group. Patients remain in PROSPECT II cohort.
- Total: Total of all reporting groups
Arm/Group | Guideline Directed Medical Therapy (GDMT) in PROSPECT-ABSORB and PROSPECT II | ABSORB BVS + GDMT in PROSPECT-ABSORB and PROSPECT II | PROSPECT II Only | Total
Number analyzed (Participants) | 89 | 93 | 716 | 898
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (9.2) | 62.0 (8.6) | 62.5 (10.4) | 62.7 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 121 | 153
  Male | 70 | 80 | 595 | 745
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 16 | 16 | 226 | 258
  Denmark | 65 | 67 | 396 | 528
  Norway | 8 | 10 | 94 | 112
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 27.3 (4.5) | 27.8 (3.8) | 27.9 (4.6) | 27.8 (4.5)
Height [Mean (Standard Deviation); unit: cm] | 174.7 (8.1) | 178.0 (7.7) | 176.2 (7.8) | 176.2 (7.8)
Weight [Mean (Standard Deviation); unit: kg] | 83.5 (16.2) | 88.0 (13.0) | 86.7 (16.3) | 86.5 (16.0)

OUTCOME MEASURES:

1. Primary Outcome: Prospect II: Patient Level Non-culprit Lesion Related Non-Culprit Major Adverse Cardiac Event (NC-MACE) Adjudicated to an Originally Untreated Non-culprit Lesion During the Entire Study Duration
Description: Patient-level rate of non-culprit lesion-related MACE (NC-MACE) evaluated at the longest follow-up available, assessed at the time when the last patient enrolled reaches at least 24 months. NC-MACE is defined as an event arising from an originally untreated NC lesion consisting of the composite of 1) cardiac death, 2) myocardial infarction, 3) unstable angina, or 4) progressive angina or anginal equivalent symptoms either 4a) requiring revascularization by coronary artery bypass grafting (CABG) or percutaneous coronary intervention (PCI), and/or 4b) with angiographic core lab-confirmed rapid lesion progression.(NC-MACE).
Time Frame: Median follow-up of 3.7 (first quartile, third quartile; 3.0, 4.4) years
Measure: Count of Participants; unit: Participants
Groups:
- Guideline Directed Medical Therapy (GDMT) in PROSPECT-ABSORB and PROSPECT II: Patient were enrolled in PROSPECT-ABSORB and randomized to GDMT group. Patients remain in PROSPECT II cohort.
- ABSORB + GDMT in PROSPECT-ABSORB and PROSPECT II: Patients were enrolled in PROSPECT-ABSORB and randomized to ABSORB + BVS + GDMT group. Patients remain in PROSPECT II cohort.
Arm/Group | Guideline Directed Medical Therapy (GDMT) in PROSPECT-ABSORB and PROSPECT II | ABSORB + GDMT in PROSPECT-ABSORB and PROSPECT II | PROSPECT II Only
Number analyzed (Participants) | 89 | 93 | 716
Participants | 15 | 10 | 41

2. Primary Outcome: Prospect Absorb: The Minimum Luminal Area (MLA) at the Randomized Non-culprit Lesion Site in Patients Treated With the ABSORB BVS + GDMT Compared to GDMT Only Measured at 25 Months
Description: The MLA at the randomized non-culprit lesion site in patients treated with Absorb BVS + GDMT compared to GDMT only as measured at 25 months.
Time Frame: 25 month
Population: Intention to treat population, defined as patients randomized to each arm and completing 25-month imaging follow-up and analyzable intravascular ultrasound (IVUS) image available
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Guideline Directed Medical Therapy | ABSORB BVS + Guideline Directed Medical Therapy
Number analyzed (Participants) | 72 | 84
mm^2 | 3.0 (1.0) | 6.9 (2.6)

ADVERSE EVENTS:
Time Frame: The entire study duration, median follow-up 3.7 (first quartile, third quartile; 3.0, 4.4) years
Description: The primary endpoint of PROSPECT II study was measured in the overall PROSPECT II cohort. As a subset of PROSPECT II, 182 patients were enrolled in PROSPECT-ABSORB and randomized to GDMT vs GDMT-ABSORB. Thus, adverse event has been shown for overall PROSPECT II cohort.
Groups:
- Guideline Directed Medical Therapy in PROSPECT-ABSORB and PROSPECT II: Patients were enrolled in PROSPECT-ABSORB and randomized to GDMT group. Patients remain in PROSPECT II cohort.
Arm/Group | Guideline Directed Medical Therapy in PROSPECT-ABSORB and PROSPECT II | ABSORB BVS + GDMT in PROSPECT-ABSORB and PROSPECT II | PROSPECT II Only
All-Cause Mortality (participants affected / at risk) | 0/89 | 2/93 | 16/716
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/93 | 2/716
Other Adverse Events (participants affected / at risk) | 0/89 | 0/93 | 0/716
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guideline Directed Medical Therapy in PROSPECT-ABSORB and PROSPECT II (N=89) | ABSORB BVS + GDMT in PROSPECT-ABSORB and PROSPECT II (N=93) | PROSPECT II Only (N=716)
Intravascular imaging related major complications requiring treatment (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) — Defined as imaging-related death or vessel dissection, perforation, spasm, or other events requiring percutaneous or surgical treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/65/NCT02171065/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/65/NCT02171065/SAP_001.pdf